

# Statistical Analysis Plan

NCT Number: NCT05341115

Title: An Open label, Multicenter, Single-arm and Prospective Study to Assess the Efficacy and Safety of Leuprorelin 3M in the Treatment of central precocious puberty (CPP)

Study Number: Leuprorelin-4002

Document Version and Date: Version 3.0, 28 May 2025

Certain information within this document has been redacted (ie, specific content is masked irreversibly from view) to protect either personally identifiable information or company confidential information.

# Statistical Analysis Plan

An Open label, Multicenter, Single-arm and Prospective Study to Assess the Efficacy and Safety of Leuprorelin 3M in the Treatment of CPP

SAP Version V3.0 May 28, 2025

For non-commercial use only

Sponsor: Takeda (China) International Trading Co., Ltd.

Project period: December, 2021 to April, 2025

Statistical analysis: LinkDoc Technology (Beijing) Co., Ltd.

#### **Statement**

The statistical analysis plan is prepared in accordance with ICH-E9 (Statistical Principles for Clinical Trials), the relevant regulations of the National Medical Products Administration (NMPA), and the standard operating procedure of LinkDoc Technology (Beijing) Co., Ltd. And it is refined based on the principles of statistical analysis in the study protocol. The mock shell (including the examples of statistical analysis tables, figures and listings) will be presented as separate documents.

For non-commercial use only

# **Approval Page**

This document has been reviewed and approved as the statistical analysis plan for this study. This document shall enter into force on the date of the last signature.

| Author: | | |
|---|---|---|
| LinkDoc Technology (Beijing) Co.,<br>Ltd. | Signature | Date<br>[DD-MM-YYYY] |
| Reviewed by: | 4 | |
| LinkDoc Technology (Beijing) Co.,<br>Ltd. | Signature | Date<br>[DD-MM-YYYY] |
| LinkDoc Technology (Beijing) Co.,<br>Ltd. | Signature | Date [DD-MM-YYYY] |
| LinkDoc Technology (Beijing) Co., Ltd. | Signature | Date [DD-MM-YYYY] |
| Takeda (China) International Trading Co., Ltd. Statistician | Signature | Date<br>[DD-MM-YYYY] |
| Takeda (China) International Trading<br>Co., Ltd.<br>Medical advisor | Signature | Date [DD-MM-YYYY] |
| Takeda (China) International Trading Co., Ltd. | Signature | Date [DD-MM-YYYY] |

# **Table of Contents**

| List of Abbreviations and Terms | 1 |
|---|---|
| 1 Study Objectives | 2 |
| 1.1 Primary Objectives | 2 |
| 1.2 Secondary Objectives | 2 |
| 2 Study Design | 2 |
| 2.1 Overall Design | 2 |
| 2.2 Study Population | 3 |
| 2.2.1 Inclusion Criterion | 3 |
| 2.2.2 Exclusion Criteria | 4 |
| 2.3 Sample Size | 5 |
| 2.4 Study Drug and Administration Method | 5 |
| Excluded Medications, Procedures, and Treatments Subject Termination or Premature Withdrawal from the Study | 5 |
| 2.6 Subject Termination or Premature Withdrawal from the Study | 5 |
| 3 Endpoint | 6 |
| 2.6 Subject Termination or Premature Withdrawal from the Study 3 Endpoint 3.1 Primary Endpoints 3.2 Secondary Endpoints 3.3 Description of Relevant Definitions 4 Analysis Set 5 Statistical Analysis | 6 |
| 3.2 Secondary Endpoints | 6 |
| 3.3 Description of Relevant Definitions | 8 |
| 4 Analysis Set | 8 |
| 5 Statistical Analysis | 9 |
| 5.1 General Principles | 9 |
| 5.2 Subject Disposition | 9 |
| 5.3 Baseline Characteristics of Subjects | 9 |
| 5.4 Drug Exposure | 11 |
| 5.5 Concomitant Treatment | 12 |
| 5.6 Primary Study Endpoint | 12 |
| 5.7 Secondary Study Endpoint | |
| 5.8 Analysis of other Variables | |
| 5.9 Discontinuation Analysis | 16 |
| 5.10 Additional Analysis | 16 |
| 5.11 Handling of Missing Values and Outliers | |
| 5.12 Interim Analysis | |
| 5.13 Explanation of Inconsistency with the Protocol | 17 |

For non-commercial use only

# **List of Abbreviations and Terms**

| Abbreviations or terminology | Explanation |
|---|---|
| AE | Adverse Event |
| AESI | Adverse Events of Special Interest |
| ALT | Alanine aminotransferase |
| AST | Aspartate aminotransferase |
| ATC | Anatomical Therapeutic Chemical Classification |
| BA/CA | Bone age/Chronological age |
| BMI | Body Mass Index |
| CI | Confidence Interval |
| CPP | Central Precocious Puberty |
| CRF | Case Report Form |
| CTCAE | Common Terminology Criteria for Adverse Events |
| FMV | First Morning Void |
| FSH | Follicle Stimulating Hormone |
| GnRH | Gonadotropin-releasing Hormone |
| GnRHa | Gonadotropin-releasing Hormone Analogs |
| hCG | Human Chorionic Gonadotropin |
| HPGA | Hypothalamic-pituitary-gonadal-axis Function |
| IRB | Institutional Review Board |
| IEC | Independent Ethics Committee |
| ITT | Intention-To-Treat (enrolled analysis population) |
| LFT | Liver Function Test |
| LH | Luteinizing Hormone |
| MedDRA | Medical Dictionary for Regulatory Activities |
| PT | Preferred Term |
| PTE | Pre-treatment Events |
| SAP | Statistical Analysis Plan |
| SAE | Serious Adverse Event |
| SAS | Statistical Analysis System |
| SOC | System Organ Class |
| SS | Safety Analysis Set (Safety Analysis Population) |
| TEAE | Treatment-Emergent Adverse Event |
| ULN | Upper Limit of Normal |
| WHODRUG | WHODrug Dictionaries |

# 1 Study Objectives

# 1.1 Primary Objectives

• To evaluate the efficacy of leuprorelin acetate depot 11.25mg 3M in subjects with CPP.

# 1.2 Secondary Objectives

• To evaluate the safety and efficacy of leuprorelin acetate depot 11.25mg 3M in subjects with CPP.

## 2 Study Design

## 2.1 Overall Design

This is an open-label, multicenter, single-arm and prospective study, to investigate the efficacy and safety of leuprolide acetate depot 11.25mg 3M formulations for the treatment of CPP in children in China. Approximately 80 subjects will be enrolled. The study includes a screening period (up to 2 weeks), a 6-month treatment period (24 weeks), and a post-treatment follow-up period (12 weeks).

The subjects will receive an injection of leuprorelin acetate depot 11.25mg 3M every 12 weeks. Pharmacokinetic studies in adults demonstrated that the quarterly formulation of 11.25 mg Leuprorelin is steadily released over 12 weeks period [3]. Each dose of the drug will be administered in outpatient hospital setting by appropriate site staff and the date of each administration will be registered on the clinical record of each child. Parents/ legal guardians of patients will be actively contacted some days before the injections to ensure them to follow the administration protocol.

Patients will be received an s.c. injection of study drug at V1, V2, V3. GnRHa stimulation will be repeated at screening visit and V2, V3 (before every s.c. injection of study drug) or at early termination. Basal LH and FSH level testing (gonadotropins and sex steroids) will be repeated at screening visit and V2, V3, V4 (before every s.c. injection of study drug) or at early termination. In this study, height and weight measurement will be performed at screening visit and V1, V2, V3, V4 (before every s.c. injection of study drug) or at early termination. Physical exams and pubertal staging will be performed at screening visit and V1, V2, V3, V4 (before every s.c. injection of study drug) or at early termination. And a BA x-ray will be taken once at the screening visit, as well as V2, V3, and V4 (before every s.c. injection of the study drug), or at early termination; the Gn in the first morning void (FMV) will be tested at the screening visit, as well as V1, V2, V3, and V4 (before each s.c. injection of the study drug), or at early termination. Adverse events will be collected and reported in this study at each study visit or at early termination, and treatment-emergent adverse events will be coded using the Medical Dictionary for Regulatory Activities (MedDRA).

V4/ET visit V 1 V3 EOS First dose Last dose Screening Follow-up Treatment period period period 24 Wks 2 Wks 12 Wks Visit 2 D -14 to D -Wk 0, 12, 24 Wk 36

Figure 2-1-1 Schematic of Study Design

V = Visit, D = Day Wk = Week, SV = Screening Visit, EOS = End of Study, ET = Early Termination

# 2.2 Study Population

The subject population in this study will be the children diagnosed with CPP who develop secondary sexual characteristics before the age of 8 years in girls or before the age of 9 years in boys.

Only those who meet all of the following inclusion criteria and none of the exclusion criteria will be eligible for the enrollment.

#### 2.2.1 Inclusion Criterion

For inclusion in the study, the subjects had to fulfill all of the following criteria:

- 1. In the opinion of the investigator, the subject and/or parent(s) or legal guardian are capable of understanding and complying with protocol requirements.
- 2. The subject or the subject's parent(s) or legally acceptable representative signs and dates a written, informed consent form and any required privacy authorization prior to the initiation of any study procedures.;
- 3. Early appearance of secondary sexual characteristics: Girls ≤8 years, Boys≤9 years;
- 4. Body weight  $\geq 20 \text{ kg}$ ;
- 5. According to the National Consensus Statement in China (2015), CPP is diagnosed when secondary sexual characteristics appeared before the age of 8 years in girls and 9 years in boys, a peak LH level > 5.0 IU/L with LH/FSH > 0.6 in stimulating test; evidence of gonadal development by ultrasonography (multiple ovarian follicles  $\geq$  4 mm in any ovary or uterine enlargement in females or testicular volume  $\geq$  4 mL in males); advanced BA  $\geq$  1 year; linear growth acceleration with higher GV than normal children. BA is determined by Greulich and Pyle standards or Tanner-Whitehouse 3 (TW3) standards at screening.

6. A male subject who is nonsterilized and sexually active with a female partner of childbearing potential agrees to use adequate contraception from signing of informed consent throughout the duration of the study and for 90 days after last dose.

- 7. A female subject of childbearing potential who is sexually active with a nonsterilized male partner agrees to use routinely adequate contraception from signing of informed consent throughout the duration of the study and for 90 days after last dose of study medication.
- 8. The female subject who, at the discretion of the investigator, is deemed to be of child bearing potential must provide negative urine pregnancy test prior to receiving any dose of study medication drug administration and negative serum hCG pregnancy test at Screening.

#### 2.2.2 Exclusion Criteria

Those who meet any of the following criteria will be excluded from this study:

- 1. The subject has received any investigational compound within 30 days prior to Screening
- 2. The subject has received GnRHa treatment in a previous clinical study or as a therapeutic agent;
- 3. The subject is an immediate family member, study site employee, or is in a dependant relationship with a study site employee who is involved in the conduct of this study (eg, spouse, parent, child, sibling) or may consent under duress;
- 4. The subject has any findings in his/her medical history, physical examination, or safety clinical laboratory tests giving reasonable suspicion of underlying disease that might interfere with the conduct of the trial;
- 5. The subject has any concomitant medical condition that, in the opinion of the investigator, may expose a subject to an unacceptable level of safety risk or that affects subject compliance;
- 6. The subject has any screening abnormal laboratory value that suggests a clinically significant underlying disease or condition that may prevent the subject from entering the study; or the subject has: creatinine ≥1.5 mg/dL, alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) 2 times the upper limit of normal (ULN), or total bilirubin 2.0 mg/dL, with AST/ALT elevated above the limits of normal values;
- 7. The subject has a history or clinical manifestations of significant adrenal or thyroid diseases or intracranial tumor OR has a history of malignant disease;
- 8. The subject has a history of hypersensitivity or allergies to leuprorelin, or related compounds including any excipients of the compound;
- 9. The subject has a diagnosis of peripheral precocious puberty;
- 10. The subject has a history of drug abuse (defined as any illicit drug use) or a history of alcohol abuse within 1 year prior to the Screening Visit;
- 11. Subject or parent(s), at the discretion of the investigator, is unlikely to comply with the protocol or is unsuitable for any of other reason;
- 12. If female, the subject is pregnant, breastfeeding, or planning to become pregnant before, during, or within 1 month after the end of the study; or planning to donate ovums during this period;

13. If male, the subject intends to donate sperm during the course of this study or for 90 days thereafter;

# 2.3 Sample Size

The calculated sample size of 70, 58, 44 and 29 was based on the assumption that the proportion of LH peak value suppression with GnRH stimulation is 80%, 85%, 90% and 95% respectively and a two-sided 95% confidence interval (CI) with a precision width of 0.2. Since the actual proportion of LH peak value suppression with GnRH stimulation in Chinese remains unknown, a conservative sample size of 70 was determined. Considering the drop-out rate 10% - 15%, a total number of 80 subjects are planned to be enrolled. This study encourages sites to enroll subjects competitively, and each site enrolls at least  $15 \sim 25$  subjects. Within each site, eligible subjects will be enrolled until the site's subject quota has been reached.

# 2.4 Study Drug and Administration Method

The study drug for this study is leuprorelin acetate depot 11.25mg 3M. The administration method is as follows: CPP subjects with body weight  $\geq$ 20 kg will receive the recommended dose of leuprorelin acetate depot 11.25 mg subcutaneous administration (SC) every 12 weeks based on the standard of  $30\sim180\mu\text{g/kg/4w}$ . It is not recommended to exceed 180  $\mu\text{g/kg}$ .

# 2.5 Excluded Medications, Procedures, and Treatments

The subjects should follow physician's instruction on Medication, Procedures and Treatments. Any concomitant medications, procedures and treatments should be recorded.

Hormonal contraceptives should be avoided during the study. In addition, all growth hormones need to be avoided for this study.

# 2.6 Subject Termination or Premature Withdrawal from the Study

The investigator may discontinue a subject's study participation at any time during the study when the subject meets the study termination criteria described in this Section. In addition, a subject may discontinue his or her participation without giving a reason at any time during the study. Should a subject's participation be discontinued, the primary reason for termination must be recorded by the investigator. In addition, efforts should be made to perform all procedures scheduled for the Early Termination Visit.

The criteria for subject termination or withdrawal are as follows:

1. Pretreatment event (PTE) or AE. The subject has experienced a PTE or AE that requires early termination because continued participation imposes an unacceptable risk to the subject's health or the subject is unwilling to continue because of the PTE or AE.

#### Liver function test (LFT) Abnormalities

Study drug should be discontinued immediately with appropriate clinical follow up (including repeat

laboratory tests, until a subject's laboratory profile has returned to normal/baseline status), if the following circumstances occur at any time during study medication treatment:

- ALT or AST  $> 8 \times ULN$ , or
- ALT or AST 5 × ULN and persists for more than 2 weeks, or
- ALT or AST  $3 \times \text{ULN}$  in conjunction with elevated total bilirubin  $2 \times \text{ULN}$  or international normalized ratio (INR) 1.5, or clinical features of jaundice
- ALT or AST 3 × ULN with appearance of fatigue, nausea, vomiting, right upper quadrant pain or tenderness, fever, rash and/or eosinophilia (5%).
- 2. Significant protocol deviation. The discovery after the first dose of study medication that the subject failed to meet protocol inclusion criterion or did not adhere to protocol requirements, and continued participation poses an unacceptable risk to the subject's health.
- 3. Lost to follow-up. The subject did not return to the clinic and attempts to contact the subject were unsuccessful. Attempts to contact the subject must be documented.
- 4. Voluntary withdrawal. The subject (or subject's legally acceptable representative) wishes to withdraw from the study. The reason for withdrawal, if provided, should be recorded in the CRF.

Note: All attempts should be made to determine the underlying reason for the withdrawal and, where possible, the primary underlying reason should be recorded (ie, withdrawal due to an AE or lack of efficacy).

- 5. Study termination. The sponsor, IRB, IEC, or regulatory agency terminates the study.
- 6. Pregnancy. The subject is found to be pregnant.

Note: If the subject is found to be pregnant, the subject must be withdrawn immediately.

- 7. Lack of efficacy. The investigator has determined that the subject is not benefiting from investigational treatment; and, continued participation would pose an unacceptable risk to the subject.
- 8. Other

#### 3 Endpoint

## 3.1 Primary Endpoints

• Percentage of subjects achieving LH peak value suppression in the GnRH stimulation test at Week 24.

Definition: The percentage of subjects with LH peak value ≤3.0 IU/L in the GnRH stimulation test at Week 24 relative to the total number of subjects in the corresponding analysis population. The LH peak value is the maximum LH value detected at 0, 30, 60 and 90 minutes after injection of the stimulation drug.

#### 3.2 Secondary Endpoints

• The percentage of subjects with Tanner stage regression or no progression at Week 24 compared with Baseline.

Definition: relative to the last available valid Tanner stage before the first administration of the leuprorelin acetate depot 11.25mg 3M, the percentage of subjects with regression or no progression in Tanner stage at Week 24 relative to the total number of subjects in the corresponding analysis population.

Progression of Tanner stage is defined as meeting any of the following conditions:

- 1) Tanner stage (left) increased compared with the baseline.
- 2) Tanner stage (right) increased compared with the baseline.
- 3) Pubic hair develops when there was none at the baseline.

No progression of Tanner stage is defined as all of the following conditions being met simultaneously:

- 1) Tanner stage (left) is the same as the baseline
- 2) Tanner stage (right) is the same as the baseline
- 3) Presence or absence of pubic hair is the same as the baseline

If Tanner stage does not meet the definition of progression, such status is classified as regression or no progression. Further, if Tanner stage meets the definition of no progression, the status is classified as no progression; if Tanner stage does not meet the definition of progression or no progression, the status is classified as regression.

• Basal LH and FSH level of subjects at Baseline, Week 24, Week 36

Definition: Basal LH and FSH values obtained from LH and FSH tests of subjects at baseline, Week 24, and Week 36.

• The percentage of subjects with decreased ratio of bone age over chronological age at Week 24 compared with Baseline.

Definition: The percentage of subjects with decreased ratio of bone age over chronological age (BA/CA) at Week 24 compared with the Baseline relative to the total number of subjects in the corresponding analysis population.

- Decrease in first morning voided (FMV) urinary Gn at Week 24 compared with Baseline.
- 1) The percentage of subjects with decreased ratio of urinary LH level in the first morning void (FMV) urinary Gn test at Week 24 compared with the Baseline.

Definition: The percentage of subjects with decreased ratio of urinary LH level in the first morning void (FMV) urinary Gn test at Week 24 among the total number of subjects in the corresponding analysis population, relative to the last available valid urinary LH level before the first administration of the leuprorelin acetate depot 11.25mg 3M.

2) The percentage of subjects with decreased ratio of urinary FSH level in the first morning void (FMV) urinary Gn test at Week 24 compared with the baseline.

Definition: The percentage of subjects with decreased ratio of urinary FSH level in the first morning void (FMV) urinary Gn test at Week 24 among the total number of subjects in the corresponding analysis population, relative to the last available valid urinary FSH level before the first administration of the leuprorelin acetate depot 11.25mg 3M.

• Incidence of treatment-emergent adverse events (TEAEs)

Definition: The percentage of subjects who experience any treatment-emergent adverse event after the first use of the study drug relative to the total number of subjects in the corresponding analysis

population. A TEAE refers to an untoward medical occurrence that occurs in a subject from the first administration of the study drug to 12 weeks after the last administration; such event is not necessarily causally related to the treatment.

#### 3.3 Description of Relevant Definitions

#### Baseline definition

For basic demographic characteristics (age, gender, ethnicity), bone age, BA/CA, predicted adult height, GnRH stimulation test (LH peak value, FSH peak value), LH and FSH (basal LH value, basal FSH value), the results from the screening visit will be taken as baseline values;

For height and weight, BMI, growth rate, estradiol/testosterone, gonads ultrasonography, pubertal stage, first morning void (FMV) urinary Gn (urinary LH value, urinary FSH value), the last available valid measurement prior to the first administration of the leuprorelin acetate depot 11.25mg 3M will be used as the baseline values.

## 4 Analysis Set

The analysis populations for this study include the enrolled analysis population, the safety analysis population, and the termination analysis population.

# **Enrolled Population:**

All eligible subjects enrolled in this study, i.e., all subjects enrolled in this study who meet the inclusion criteria and do not meet any of the exclusion criteria, regardless of whether they receive the study drug, will be included in this analysis set. Unless otherwise specified, the primary and secondary study endpoints (except for adverse event analysis), and baseline characteristics of subjects will be analyzed based on the enrolled population.

For the subjects with significant protocol deviation in this population, the final decision on whether the data affected by the significant protocol deviation is included in the final analysis will be determined at the data review meeting.

#### **Safety Population:**

All included patients who have been under treatment with Leuprorelin or who are first prescribed Leuprorelin, receive at least one dose and complete one follow-up visit. A supplementary analysis of the primary study endpoints will be performed based on the safety population as per the actual data of the safety population. The analysis of drug exposure, adverse events and concomitant medications will be based on the safety population.

Completion of one follow-up is defined as subjects with at least one post-baseline data available. Post-baseline data include the results of the following examinations: vital signs, growth rate, weight, height, BMI, concomitant medications, Tanner stage assessment, gonads ultrasonography, bone age, BA/CA, hematology, urinalysis, clinical chemistry, contraceptive consultation (if applicable), electrocardiogram, estradiol or testosterone, FMV urinary Gn, stimulation test, basal LH and FSH, AE assessment, PTE, physical examination, concomitant non-drug therapy, etc.

#### **Discontinuation population:**

Patients who discontinue the use of Leuprorelin, are lost to follow-up, withdraw from the study or are dead. Discontinuation analysis will be based on the discontinuation population.

# **5 Statistical Analysis**

# 5.1 General Principles

Descriptive analyses are the primary focus of this study and no preplanned hypothesis testing will be performed.

All statistical analyses will be programmed and calculated by SAS 9.4 statistical analysis software.

Continuous indicators will be described by number of cases (missing numbers), arithmetic mean, standard deviation, median, 25th and 75th percentile, minimum and maximum; discrete indicators will be described by number of cases and percentages, with a 95% confidence interval if necessary;

Unless otherwise specified, all statistical analysis results will be presented by gender group.

Unless otherwise specified, all missing data will not be imputed.

In this study, MedDRA\_28\_0\_Chinese and WHO\_DD\_V3.02\_2025-06\_Chinese coding dictionaries (version numbers will be adjusted based on actual conditions) will be used to code relevant medical events and drugs used.

# **5.2 Subject Disposition**

Describe the distribution of all screened and included patients in the study, including the number of screened subjects, the number and percentage of subjects who failed screening, the reason and percentage of screening failure, the number and percentage of included patients, the number and percentage of subjects with early termination of treatment, the reason and percentage of early termination of treatment, the number and percentage of subjects with study termination, the reason and percentage of study termination, the number and percentage of subjects with protocol deviation, the number and percentage of subjects with different types of protocol deviation, and the number of different types of protocol deviation.

Describe the distribution of subjects in each analysis set, including the number of subjects in each analysis set (including the enrolled population, safety population, and discontinuation population); describe the number and percentage of subjects enrolled at each site; list the excluded subjects in the enrolled population and safety population (including subject number, age, gender, reason for exclusion, etc.); list subjects with protocol deviations (including subject number, age, gender, severity, protocol deviation type, and specific description).

#### 5.3 Baseline Characteristics of Subjects

The description of baseline characteristics will be based on the enrolled population.

The basic information of baseline characteristics of subjects will be described according to general

principles, mainly including:

• Baseline demographics: age, gender, ethnicity, height, weight, body mass index (BMI), bone age, BA/CA, predicted adult height, growth rate; Where BMI=weight (kg)/height (m)<sup>2</sup>, BMI can be described in sections according to WHO classification criteria (based on different ages, BMI grade is divided into severely thinness, thinness, normal, overweight and obesity). The criteria C is summarized as follows, corresponding to age:

♦ Severe thinness: BMI<-3SD;</p>

♦ Thinness: -3SD≤BMI<-2SD;</p>

♦ Normal: -2SD≤BMI≤1SD;

♦ Overweight: 1SD<BMI≤2SD;

 $\Leftrightarrow$  Obesity: 2SD  $\leq$  BMI, see Appendix A [1] for specific classification criteria.

The demographic data of subjects will be presented in listings.

• Prior medical history and concomitant diseases/pre-treatment events: presence or absence of prior medical history, name of medical history, presence or absence of concomitant diseases/pre-treatment events, name of disease/pre-treatment events. The names of disease/pre-treatment event will be presented in the form of SOC (System Organ Class) and PT (Preferred Term). The prior medical history and a list of concomitant diseases/pre-treatment events of the subjects will be presented in listings.

The prior medical history refers to any significant condition or disease related to the disease under study that has recovered at or prior to signing informed consent, and any significant condition or disease related to the disease under study that has healed within 1 year prior to signing informed consent; concomitant disease refers to is a significant condition or disease that is still present at the time of signing the informed consent form, including clinically significant abnormal laboratory values, electrocardiogram, or physical examination abnormalities at screening; a pre-treatment event refers to all untoward medical occurrences that occur in the subjects who have signed the informed consent to participate in the study before the use of any study drug.

• Prior medication history: presence or absence of medication history, names of drugs. Specific drugs will be summarized and analyzed according to ATC therapeutic classification categories (ATC-2) and Preferred Names. A list of prior medication history list for subjects will be presented in listings.

The prior medication is any medication related to eligibility criteria that has been discontinued at or within 1 month prior to signing informed consent.

- Information on estradiol/testosterone tests at baseline: presence or absence of estradiol test, quantitative test results for estradiol, qualitative test results for estradiol, presence or absence of testosterone test, quantitative test results for testosterone, qualitative test results for testosterone.
- Results of gonadal ultrasound examinations at baseline: For females, describe pelvic ultrasound information, including presence or absence of pelvic ultrasound, the volume of the left ovary, the volume of the right ovary, uterine size, follicle volume, number of follicles; for males, describe presence or absence of gonadal ultrasound, the left testicular volume, and the right testicular volume.
- GnRH stimulation LH peak value, GnRH stimulation FSH peak value, LH peak value/FSH

peak value during the subject's baseline period.

• Pubertal staging (i.e., Tanner staging) of subjects at baseline: presence or absence of Tanner staging assessment, Tanner stage (left), Tanner stage (right), and presence or absence of pubic hair.

# 5.4 Drug Exposure

Drug exposure will be summarized by treatment duration of leuprolide based on the enrolled population. The duration of treatment with leuprolide is defined as the time interval from the first injection of leuprolide to the last injection of leuprolide in the subjects. The overdose of leuprolide will also be summarized.

The use of leuprolide will be described in accordance with general principles, Including: duration of treatment, duration of drug exposure, actual number of leuprorelin injections, whether the first injection of leuprorelin is received, whether the second injection of leuprorelin is received, whether the third injection of leuprorelin is received, actual dose administered for the first injection ( $\mu g/kg/4w$ ), intended dose for the first injection ( $\mu g/kg/4w$ ), actual dose administered for the second injection ( $\mu g/kg/4w$ ), intended dose for the second injection ( $\mu g/kg/4w$ ), actual dose administered for the third injection ( $\mu g/kg/4w$ ), average actual dose administered ( $\mu g/kg/4w$ ), average intended dose ( $\mu g/kg/4w$ ), cumulative actual dose administered ( $\mu g/kg/4w$ ), number of times for the actual dose in subjects exceeding 180  $\mu g/kg/4w$ , number of times for the intended dose in subject exceeding 180  $\mu g/kg/4w$ , and relative dose intensity. The relevant definitions or calculation formulas are as follows:

- 1) Duration of treatment (days) = date of last injection of leuprorelin for the subject date of first injection of leuprorelin for the subject + 1;
- 2) Duration of drug exposure (days) = date of last injection of leuprorelin for the subject date of first injection of leuprorelin for the subject + 84;
- 3) The mean actual dose administered (ug/kg/4w) is equal to the mean of the actual dose administered (ug/kg/4w) of all non-missing injections of leuprolide for the subject;
- 4) The mean intended dose (ug/kg/4w) is equal to the mean of all non-missing intended doses of leuprolide injections (ug/kg/4w) for the subject;
- 5) Cumulative actual dose administered (mg) is equal to the sum of all non-missing actual doses of leuprolide injections (mg) for the subject;
- 6) Cumulative intended dose (mg) is equal to the sum of all non-missing intended doses of leuprorelin injections (mg) for the subject;
- 7) Relative dose intensity = [Cumulative actual dose administered (mg) / Cumulative intended dose (mg)] × 100%;
- 8) Intended dose (ug/kg/4w) = Intended dose (ug/kg) / 3 = [Intended dose (mg)  $\times$  1000 / Body weight (kg)] / 3;
- 9) Actual dose administered (ug/kg/4w) = Actual dose administered (ug/kg)/actual time interval (4w) from current injection to the next injection of leuprolide (4w) = [actual dose administered (mg)\*1000/body weight (kg)]/[(date of next injection date of current injection)/28. If there is no next injection, fill in the actual time interval with three 4Ws;

Overdose of leuprolide will be described in accordance with general principles, including presence

or absence of overdose, number of overdose occurrences, presence or absence of related AE, preferred term for related AE, causes for overdose. The relevant definitions or calculation formulas are as follows:

- 10) Leuprolide overdose is defined as a situation where the subject intentionally or accidentally receives a dose of leuprolide that exceeds the dose assigned to the subject in the study protocol;
- 11) The number of overdose occurrences is equal to the number of "Yes" recorded for "Whether the study drug is overdosed" in all drug overdose records.

The administration of leuprolide to the subjects is present in listings.

#### **5.5** Concomitant Treatment

The concomitant medications and concomitant non-drug therapies for the subjects will be described in accordance with general principles based on the safety population, Including: presence or absence of concomitant medication, name of medication, reason for medication, presence or absence of concomitant non-drug therapy, reason for non-drug therapy. The same individual subject can have one or more reasons for medication/non-drug treatment, and the number and percentage of cases with different reasons for use will be counted separately. The denominator of percentage calculation will be the number of non-missing subjects in the safety population. The number and percentage of subjects using each specific drug will be summarized by ATC classification system and common terminology of World Health Organization. A list of concomitant medications and a list of concomitant non-drug therapies for subjects will be presented in listings.

Concomitant medication is defined as any drugs administered to the subject other than the study drug from the time of signing the informed consent form to the end of the study. That is, a drug is considered a concomitant medication if it meets either of the following conditions: ① The "whether it is ongoing" status is "Yes", and the start date of medication is earlier than the study completion date or study termination date; ② The "whether it is ongoing" status is "No", the start date of medication is earlier than the study completion date or study termination date, and the end date of medication is later than the date of signing the informed consent form.

Concomitant non-drug therapy is defined as any non-drug therapy received by the subject from the time of signing the informed consent form to the end of the study. That is, a therapy is considered a concomitant non-drug therapy if it meets either of the following conditions: ① The "whether it is ongoing" status is "Yes", and the start date of therapy is earlier than the study completion date or study termination date; ② The "whether it is ongoing" status is "No", the start date of therapy is earlier than the study completion date or study termination date, and the end date of therapy is later than the date of signing the informed consent form.

# **5.6 Primary Study Endpoint**

The analysis of the primary study endpoint will be based on the enrolled population.

Describe the number and percentage of subjects achieving LH peak value suppression in the GnRH stimulation test at Week 12 and Week 24, and estimate their 95% confidence interval using Clopper-pearson method. A subject is considered not to achieve LH peak value suppression if the LH peak value of the GnRH stimulation test at Week 12 and Week 24 is missing.

The trend of the percentage of subjects achieving LH peak value suppression in the GnRH stimulation test at Week 12 and Week 24 will be presented in figures by gender, with 95% confidence intervals

estimated by Clopper-pearson method.

The subjects' GnRH stimulation LH values by visit will be presented in listings.

A sensitivity analysis will be performed for the primary study endpoint, i.e., if a subject has missing LH peak value in the GnRH stimulation test at Week 12 and Week 24, the primary study endpoint will be analyzed after the nearest available measurement from Week 12 and Week 24 (non-baseline) is used as a missing imputation.

# 5.7 Secondary Study Endpoint

The analysis of the secondary study endpoint will be based on the enrolled population. The following descriptive analyses by gender will be performed separately for the secondary study endpoints according to the general principles:

1) The percentage of subjects with Tanner stage regression or no progression at Week 24 compared with Baseline.

Describe the number and percentage of subjects with Tanner stage regression or no progression at Week 24 compared with Baseline, and estimate the 95% confidence interval using the Clopper-Pearson method. A subject is considered to have no regression or no progression in Tanner stage if the Tanner staging result at Week 24 is missing.

The Tanner staging results by visit will be presented in listings.

A sensitivity analysis will be performed for this endpoint, i.e., if a subject has a missing Tanner staging result at Week 24, this endpoint will be analyzed after the nearest available measurement from Week 24 (non-baseline) is used as a missing imputation.

2) Basal LH and FSH level of subjects at Baseline, Week 24, Week 36

The distribution of LH and FSH test results (including basic LH levels and basic FSH levels) in subjects at Baseline, Week 24, and Week 36 will be described using the number of cases, mean, standard deviation, median, 25th and 75th percentiles, minimum and maximum values. Trend graphs of basal LH and box plots of basal FSH change trends will be plotted separately for subjects by gender at baseline, Week 24, and Week 36.

The baseline LH and FSH values for subjects by visit will be presented in listings.

A sensitivity analysis will be performed for this endpoint, i.e. if the results of basal LH and FSH tests at baseline, Week 24, or Week 36 for a subject are "<xx.xx", "xx.xx" will be used for imputation; if there are still missing values, the 0-minute results of the stimulation test during the same visit period will be used for imputation before the analysis of this indicator.

3) The percentage of subjects with decreased ratio of bone age over chronological age (BA/CA) at Week 24 compared with the Baseline.

Describe the number and percentage of subjects with decreased ratio of bone age over chronological age (BA/CA) at Week 24 compared with Baseline and estimate their 95% confidence interval using Clopper-pearson method. A subject is considered not to achieve decreased ratio of BA/CA if the BA/CA value is missing at Week 24.

The bone age/chronological age (BA/CA) results by visit will be presented in listings.

A sensitivity analysis will be performed for this endpoint, i.e., if a subject has missing BA/CA value at Week 24, this endpoint will be analyzed after the nearest available measurement from Week 24

(non-baseline) is used as a missing imputation.

4) The percentage of subjects with decrease in first morning voided (FMV) urinary Gn at Week 24 compared with Baseline.

Describe the number and percentage of subjects with decreased urinary LH and decreased urinary FSH values in the urinary Gn test results of the first morning void (FMV) at Week 24 compared with Baseline, separately, and estimate their 95% confidence intervals using Clopper-pearson method.

For urinary LH and FSH values in urinary Gn test results of the first morning void (FMV) at Baseline and Week 24, any value that is <0.05 should be recorded as "<0.05". If both the Baseline and Week 24 results are "<0.05", the assessment of such decrease will be treated as missing. If there is at most one "<0.05" result, a comparison can be performed. See Appendix B for the reasons of above processing.

If a subject has a missing value for an indicator in the urinary Gn test results of the first morning void (FMV) at Baseline or Week 24, the subject will be considered not to achieve a decrease in that indicator of the FMV urinary Gn.

The urinary Gn test results of the first morning void (FMV) for the subjects by visit will be presented in listings.

Two sensitivity analyses will be conducted separately for each of the two indicators of this endpoint. For the first sensitivity analysis, if a subject has a missing value for an indicator in urinary Gn test results of the first morning void (FMV) at Week 24, this indicator will be analyzed after the nearest available measurement from Week 24 (non-baseline) is used as a missing imputation. Sensitivity analysis will be performed using the Gn results of the first morning void (FMV) collected by EDC directly for the second time. If the urinary Gn test results of the first morning void (FMV) for the subject at Baseline or week 24 were missing, it was considered that he/she did not achieve a decrease in that indicator of the FMV urinary Gn.

5) Incidence of treatment-emergent adverse events (TEAEs)

The analysis of adverse events will be based on the safety population. The number of cases, number of occurrences, and incidence of TEAEs will be analyzed. All adverse events will be coded using MedDRA 28 0 Chinese (the version number will be adjusted based on the actual situation).

The number of cases, number of occurrences and incidence of all AEs, TEAEs, SAEs, adverse events of special interest (AESIs), AEs leading to discontinuation, AEs leading to dose interruption, AEs leading to dose reduction, AEs related to study drug, AEs leading to trial withdrawal, AEs leading to death, AEs leading to death, and AEs with Grade 3 and above will be summarized separately.

Relevant characteristic information of adverse events will be described, including: severity (i.e., CTCAE grade), outcome, causal relationship with the study drug leuprolide, relationship with study procedures, and frequency of occurrence.

The distribution of all AEs, TEAEs, SAEs, AESIs, AEs leading to discontinuation, AEs leading to dose interruption, AEs leading to dose reduction, AEs with Grade 3 and above, AEs related to the study drug, AEs leading to trial withdrawal, and AEs leading to death will be summarized according to the SOC and PT in the MedDRA coding system.

The lists of adverse events, adverse events related to the study drug and serious adverse events will be presented listings.

The relevant definitions of adverse events are as follows:

An adverse event (AE) is defined as any untoward medical occurrence in a clinical investigation subject first administered a drug

A treatment-emergent adverse event (TEAE) is an untoward medical occurrence that occurs in a subject from the first administration of the study drug to 12 weeks after the last administration of the study drug; it does not necessarily have to have a causal relationship with this treatment.

A serious adverse event (SAE) is any untoward medical occurrence occurring at any dose level that meets one of the following criteria: a. results in death; b. life-threatening; c. requirements for hospitalization or prolongation of hospitalization; d. results in permanent or significant disability/incapacity; e. leads to a congenital anomaly/birth defect.; f. Is an important medical event that satisfies any of the following: 1. May require intervention to prevent items a through e above; 2. May expose the subject to danger, even though the event is not immediately life threatening or fatal or does not result in hospitalization.

Adverse events of special interest (AESIs) are scientific and medical events specifically related to the product or study: a. injection site reactions, b. emotional instability, c. hypersensitivity, d. convulsions, e. slipped capital femoral epiphysis.

Adverse events leading to discontinuation will be defined as specific AEs leading to discontinuation of the study drug Leuprorelin acetate depot 11.25mg 3M.

Adverse events leading to dose interruption will be defined as specific AEs that result in the interruption of the use of study drug Leuprorelin acetate depot 11.25mg 3M.

Adverse events leading to dose reduction will be defined as specific AEs that result in the dose reduction of the study drug Leuprorelin acetate depot 11.25mg 3M.

Adverse events related to the study drug are the specific adverse events that are causally related to the study drug Leuprorelin acetate depot 11.25mg 3M.

## 5.8 Analysis of other Variables

Other indicators will be analyzed based on the enrolled population. The following descriptive analyses of estradiol and testosterone by gender will be performed according to the general principles:

The distribution of estradiol/testosterone test results (including quantitative results of estradiol tests, quantitative results of testosterone tests, and qualitative results of testosterone tests) in subjects at Baseline, Week 12, Week 24, and Week 36 will be described using the number of cases, mean, standard deviation, median, 25th and 75th percentiles, minimum and maximum. Additionally, the differences between the quantitative results of estradiol/testosterone tests at Week 12, Week 24, and Week 36 and those at baseline will be described separately; contingency tables will be used to describe the changes in the qualitative results of estradiol/testosterone tests at Week 12, Week 24, and Week 36 compared with Baseline.

The list of estradiol/testosterone results by visit will be presented in listing.

#### 5.9 Discontinuation Analysis

The discontinuation analysis will be based on the discontinuation population. The number and percentage of subjects whose study termination is caused by adverse events, death, or other reasons will be calculated separately, and the tolerability of leuprolide will be evaluated through the termination rate.

# 5.10 Additional Analysis

The following supplemental analyses will be performed to assess the robustness of the study results.

- 1) Conduct two supplementary analyses for the primary study endpoint: i. In the enrolled population, the analysis will be based on the non-missing data, i.e. if the LH peak value values of the GnRH stimulation test at Week 12 and Week 24 are missing, the results will be considered as unknown and will not be included in the denominator for calculating the percentage, and then the primary study endpoint will be analyzed. The analysis method is the same as that in Section 5.6; ii. The primary study endpoint will be analyzed based on the safety population, if applicable.
- 2) Supplemental analyses will be performed on the enrolled population for the following three secondary study endpoints:
  - The percentage of subjects with Tanner stage regression or no progression at Week 24 compared with Baseline
  - The percentage of subjects with decreased ratio of bone age over chronological age at Week 24 compared with Baseline
  - The percentage of subjects with a decrease in Gn of the first morning void (FMV) at Week 24 compared with the baseline (For the Gn results of the first morning void at Baseline and Week 24, re-processed data will be used, see Part 4) in Section 5.7).

The analysis will be conducted based on non-missing data. Specifically, if a subject has missing data for a secondary study endpoint at Week 24, the result will be regarded as unknown and will not be included in the denominator for percentage calculation. The secondary study endpoint will then be analyzed using the same method as described in Section 5.7.

#### 5.11 Handling of Missing Values and Outliers

For time variables involved in the analysis that require imputation: if the year is missing, no imputation will be performed; if the month is missing and median imputation (06/30) does not cause logical issues, median imputation will be adopted, and if there is a logical issue, the handling will be determined based on specific circumstances; if the day is missing and median imputation (15) does not cause logical issues, median imputation will be used; if logical issues arise, the handling will depend on the specific situation.

For the imputation of the occurrence date of an adverse event (AE) (if needed), it will be performed in a way that maximizes the chance of the event being classified as a treatment-emergent adverse

event (TEAE). Specifically: if the year is missing, directly impute the first leuprolide injection date; if the month is missing and the occurrence year matches the year of the first leuprolide injection date, impute the first leuprolide injection date; if the month is missing and the occurrence year differs from the year of first leuprolide injection date, then impute the first day of the occurrence year; if the day is missing and the year and month of occurrence match those of the first leuprolide injection date, impute first leuprolide injection date; if the day is missing and the year and month of occurrence differ from those of the first leuprolide injection date, then impute as the first day of occurrence month.

Unless otherwise specified, no imputation will be performed for other data.

Whether a value is an outlier will be judged based on the actual condition of the data. Records identified as outliers will be handled accordingly after data management queries and medical review.

# 5.12 Interim Analysis

The cutoff date for data collection of the interim analysis in this study is planned as August 31, 2023.

For subjects whose primary endpoint or each secondary endpoint can be completely defined by the cutoff date of data collection for the interim analysis, the corresponding endpoints will be analyzed using the methods described in Sections 5.6 and 5.7.

For subjects whose primary endpoint or each secondary endpoint cannot be completely defined by the cutoff date of data collection for the interim analysis, relevant descriptions will be made for the available data on LH peak value in GnRH stimulation test, Tanner stage, basal LH and FSH levels, bone age/chronological age (BA/CA), Gn of first morning void (FMV), and treatment-emergent adverse events.

# 5.13 Explanation of Inconsistency with the Protocol

The contents of this SAP that are inconsistent with the protocol are summarized as follows:

- 1. The definition of the enrolled population in Section 13.5 of the protocol refers to all eligible subjects enrolled in this study, and the above definition is refined in this SAP, as shown in Section 4.
- 2. Section 13.6 of the Protocol stipulates that all analyses will be based on observed data without imputation of missing data. This SAP will perform imputation for some time variables, and the imputation rules are described in Section 5.11.

# **Appendices**

# Appendix A BMI Grading Criteria by WHO for Children Aged 5-19 years [1]

Table 6-1-3 BMI Classification Criteria for 5-19 Years Old (Male)

| Month | SD3neg | SD2neg | SD1neg | SD0 | SD1 | SD2 |
|-------|--------|--------|--------|--------|--------|--------|
| 61 | 12.118 | 13.031 | 14.071 | 15.264 | 16.645 | 18.259 |
| 62 | 12.115 | 13.027 | 14.066 | 15.262 | 16.648 | 18.273 |
| 63 | 12.114 | 13.024 | 14.063 | 15.26 | 16.653 | 18.29 |
| 64 | 12.114 | 13.022 | 14.061 | 15.26 | 16.659 | 18.308 |
| 65 | 12.114 | 13.021 | 14.06 | 15.262 | 16.667 | 18.328 |
| 66 | 12.115 | 13.021 | 14.06 | 15.264 | 16.676 | 18.35 |
| 67 | 12.117 | 13.021 | 14.061 | 15.268 | 16.686 | 18.374 |
| 68 | 12.121 | 13.023 | 14.063 | 15.274 | 16.699 | 18.399 |
| 69 | 12.125 | 13.026 | 14.067 | 15.28 | 16.712 | 18.427 |
| 70 | 12.129 | 13.03 | 14.071 | 15.288 | 16.727 | 18.456 |
| 71 | 12.135 | 13.035 | 14.077 | 15.296 | 16.743 | 18.487 |
| 72 | 12.141 | 13.04 | 14.083 | 15.306 | 16.761 | 18.52 |
| 73 | 12.148 | 13.047 | 14.09 | 15.317 | 16.78 | 18.554 |
| 74 | 12.155 | 13.053 | 14.098 | 15.328 | 16.799 | 18.589 |
| 75 | 12.163 | 13.061 | 14.107 | 15.341 | 16.82 | 18.626 |
| 76 | 12.171 | 13.069 | 14.116 | 15.354 | 16.842 | 18.665 |
| 77 | 12.18 | 13.077 | 14.126 | 15.368 | 16.864 | 18.704 |
| 78 | 12.189 | 13.086 | 14.136 | 15.382 | 16.888 | 18.745 |
| 79 | 12.198 | 13.095 | 14.147 | 15.398 | 16.913 | 18.788 |
| 80 | 12.208 | 13.105 | 14.158 | 15.414 | 16.938 | 18.831 |
| 81 | 12.218 | 13.115 | 14.17 | 15.43 | 16.964 | 18.876 |
| 82 | 12.228 | 13.126 | 14.183 | 15.447 | 16.991 | 18.922 |
| 83 | 12.239 | 13.136 | 14.195 | 15.465 | 17.019 | 18.969 |
| 84 | 12.25 | 13.148 | 14.209 | 15.483 | 17.047 | 19.017 |
| 85 | 12.261 | 13.159 | 14.222 | 15.502 | 17.076 | 19.066 |
| 86 | 12.272 | 13.171 | 14.236 | 15.521 | 17.106 | 19.116 |
| 87 | 12.283 | 13.183 | 14.25 | 15.541 | 17.136 | 19.168 |
| 88 | 12.295 | 13.195 | 14.265 | 15.561 | 17.167 | 19.22 |
| 89 | 12.307 | 13.208 | 14.28 | 15.581 | 17.199 | 19.274 |
| 90 | 12.319 | 13.221 | 14.295 | 15.602 | 17.231 | 19.328 |
| 91 | 12.331 | 13.234 | 14.311 | 15.624 | 17.264 | 19.383 |
| 92 | 12.343 | 13.247 | 14.327 | 15.646 | 17.297 | 19.44 |
| 93 | 12.356 | 13.26 | 14.343 | 15.668 | 17.331 | 19.497 |
| 94 | 12.368 | 13.274 | 14.36 | 15.69 | 17.366 | 19.555 |

| Month | SD3neg | SD2neg | SD1neg | SD0 | SD1 | SD2 |
|-------|--------|--------|--------|--------|--------|--------|
| 95 | 12.381 | 13.288 | 14.377 | 15.713 | 17.401 | 19.615 |
| 96 | 12.394 | 13.302 | 14.394 | 15.737 | 17.437 | 19.675 |
| 97 | 12.407 | 13.317 | 14.412 | 15.761 | 17.473 | 19.736 |
| 98 | 12.42 | 13.331 | 14.429 | 15.785 | 17.51 | 19.798 |
| 99 | 12.434 | 13.346 | 14.447 | 15.809 | 17.548 | 19.862 |
| 100 | 12.447 | 13.361 | 14.466 | 15.834 | 17.586 | 19.926 |
| 101 | 12.461 | 13.376 | 14.484 | 15.86 | 17.624 | 19.99 |
| 102 | 12.475 | 13.392 | 14.503 | 15.886 | 17.663 | 20.056 |
| 103 | 12.489 | 13.408 | 14.523 | 15.912 | 17.702 | 20.123 |
| 104 | 12.503 | 13.424 | 14.542 | 15.938 | 17.742 | 20.19 |
| 105 | 12.518 | 13.44 | 14.562 | 15.965 | 17.783 | 20.258 |
| 106 | 12.532 | 13.456 | 14.582 | 15.992 | 17.824 | 20.327 |
| 107 | 12.547 | 13.473 | 14.603 | 16.02 | 17.866 | 20.397 |
| 108 | 12.562 | 13.491 | 14.624 | 16.049 | 17.908 | 20.468 |
| 109 | 12.578 | 13.508 | 14.646 | 16.078 | 17.952 | 20.54 |
| 110 | 12.594 | 13.526 | 14.668 | 16.108 | 17.996 | 20.613 |
| 111 | 12.61 | 13.545 | 14.691 | 16.138 | 18.04 | 20.687 |
| 112 | 12.626 | 13.564 | 14.714 | 16.169 | 18.086 | 20.763 |
| 113 | 12.643 | 13.583 | 14.738 | 16.201 | 18.132 | 20.839 |
| 114 | 12.661 | 13.603 | 14.763 | 16.233 | 18.179 | 20.916 |
| 115 | 12.679 | 13.624 | 14.788 | 16.266 | 18.227 | 20.994 |
| 116 | 12.697 | 13.645 | 14.814 | 16.3 | 18.276 | 21.074 |
| 117 | 12.716 | 13.667 | 14.84 | 16.335 | 18.326 | 21.154 |
| 118 | 12.735 | 13.689 | 14.867 | 16.37 | 18.376 | 21.234 |
| 119 | 12.755 | 13.712 | 14.895 | 16.406 | 18.428 | 21.317 |
| 120 | 12.775 | 13.735 | 14.923 | 16.443 | 18.48 | 21.4 |
| 121 | 12.796 | 13.759 | 14.952 | 16.481 | 18.532 | 21.483 |
| 122 | 12.817 | 13.784 | 14.982 | 16.519 | 18.586 | 21.568 |
| 123 | 12.838 | 13.808 | 15.012 | 16.558 | 18.64 | 21.653 |
| 124 | 12.86 | 13.834 | 15.043 | 16.597 | 18.696 | 21.739 |
| 125 | 12.882 | 13.86 | 15.074 | 16.638 | 18.751 | 21.826 |
| 126 | 12.905 | 13.886 | 15.106 | 16.679 | 18.808 | 21.914 |
| 127 | 12.928 | 13.913 | 15.139 | 16.72 | 18.865 | 22.002 |
| 128 | 12.952 | 13.941 | 15.172 | 16.763 | 18.923 | 22.09 |
| 129 | 12.976 | 13.969 | 15.206 | 16.806 | 18.982 | 22.18 |
| 130 | 13.001 | 13.998 | 15.241 | 16.85 | 19.042 | 22.271 |
| 131 | 13.026 | 14.027 | 15.276 | 16.894 | 19.102 | 22.362 |
| 132 | 13.051 | 14.056 | 15.312 | 16.939 | 19.163 | 22.452 |
| 133 | 13.077 | 14.087 | 15.348 | 16.985 | 19.224 | 22.544 |
| 134 | 13.103 | 14.117 | 15.385 | 17.031 | 19.287 | 22.637 |

| Month | SD3neg | SD2neg | SD1neg | SD0 | SD1 | SD2 |
|-------|--------|--------|--------|----------------|--------|--------|
| 135 | 13.13 | 14.148 | 15.422 | 17.078 | 19.349 | 22.729 |
| 136 | 13.157 | 14.18 | 15.461 | 17.126 | 19.413 | 22.822 |
| 137 | 13.185 | 14.212 | 15.499 | 17.175 | 19.477 | 22.915 |
| 138 | 13.213 | 14.245 | 15.539 | 17.224 | 19.542 | 23.009 |
| 139 | 13.241 | 14.278 | 15.578 | 17.273 | 19.607 | 23.104 |
| 140 | 13.27 | 14.312 | 15.619 | 17.324 | 19.674 | 23.199 |
| 141 | 13.3 | 14.347 | 15.66 | 17.375 | 19.741 | 23.293 |
| 142 | 13.33 | 14.382 | 15.702 | 17.427 | 19.808 | 23.389 |
| 143 | 13.36 | 14.417 | 15.745 | 17.48 | 19.877 | 23.485 |
| 144 | 13.391 | 14.453 | 15.788 | 17.533 | 19.946 | 23.581 |
| 145 | 13.422 | 14.49 | 15.833 | 17.588 | 20.015 | 23.677 |
| 146 | 13.454 | 14.528 | 15.877 | 17.643 | 20.086 | 23.774 |
| 147 | 13.487 | 14.566 | 15.923 | 17.698 | 20.157 | 23.871 |
| 148 | 13.52 | 14.605 | 15.969 | 17.755 | 20.229 | 23.969 |
| 149 | 13.554 | 14.644 | 16.016 | 17.812 | 20.302 | 24.067 |
| 150 | 13.588 | 14.684 | 16.063 | 17.87 | 20.375 | 24.165 |
| 151 | 13.622 | 14.724 | 16.112 | 17.929 | 20.449 | 24.263 |
| 152 | 13.658 | 14.766 | 16.161 | 17.989 | 20.524 | 24.362 |
| 153 | 13.693 | 14.807 | 16.21 | 18.049 | 20.599 | 24.46 |
| 154 | 13.729 | 14.849 | 16.26 | <b>5</b> 18.11 | 20.675 | 24.559 |
| 155 | 13.766 | 14.892 | 16.311 | 18.171 | 20.751 | 24.658 |
| 156 | 13.802 | 14.935 | 16.362 | 18.233 | 20.829 | 24.757 |
| 157 | 13.839 | 14.979 | 16.414 | 18.296 | 20.906 | 24.856 |
| 158 | 13.877 | 15.023 | 16.466 | 18.359 | 20.984 | 24.954 |
| 159 | 13.915 | 15.067 | 16.519 | 18.422 | 21.062 | 25.053 |
| 160 | 13.953 | 15.112 | 16.572 | 18.486 | 21.14 | 25.152 |
| 161 | 13.991 | 15.157 | 16.625 | 18.55 | 21.219 | 25.249 |
| 162 | 14.029 | 15.202 | 16.679 | 18.615 | 21.298 | 25.347 |
| 163 | 14.068 | 15.247 | 16.733 | 18.68 | 21.376 | 25.444 |
| 164 | 14.107 | 15.293 | 16.787 | 18.744 | 21.455 | 25.54 |
| 165 | 14.145 | 15.338 | 16.841 | 18.81 | 21.534 | 25.635 |
| 166 | 14.184 | 15.384 | 16.895 | 18.875 | 21.613 | 25.731 |
| 167 | 14.222 | 15.429 | 16.95 | 18.94 | 21.691 | 25.825 |
| 168 | 14.261 | 15.475 | 17.004 | 19.005 | 21.77 | 25.918 |
| 169 | 14.299 | 15.521 | 17.058 | 19.07 | 21.848 | 26.011 |
| 170 | 14.337 | 15.566 | 17.113 | 19.135 | 21.926 | 26.103 |
| 171 | 14.375 | 15.611 | 17.167 | 19.2 | 22.004 | 26.194 |
| 172 | 14.414 | 15.657 | 17.221 | 19.265 | 22.081 | 26.284 |
| 173 | 14.451 | 15.702 | 17.275 | 19.329 | 22.158 | 26.373 |
| 174 | 14.489 | 15.747 | 17.329 | 19.394 | 22.235 | 26.462 |

| Month | SD3neg | SD2neg | SD1neg | SD0 | SD1 | SD2 |
|-------|--------|--------|--------|--------|--------|--------|
| 175 | 14.526 | 15.791 | 17.382 | 19.458 | 22.311 | 26.549 |
| 176 | 14.563 | 15.836 | 17.435 | 19.522 | 22.387 | 26.635 |
| 177 | 14.6 | 15.88 | 17.489 | 19.585 | 22.462 | 26.72 |
| 178 | 14.636 | 15.924 | 17.541 | 19.649 | 22.537 | 26.804 |
| 179 | 14.672 | 15.968 | 17.594 | 19.712 | 22.611 | 26.887 |
| 180 | 14.708 | 16.011 | 17.647 | 19.774 | 22.685 | 26.969 |
| 181 | 14.744 | 16.054 | 17.699 | 19.837 | 22.758 | 27.051 |
| 182 | 14.779 | 16.097 | 17.75 | 19.899 | 22.831 | 27.13 |
| 183 | 14.814 | 16.14 | 17.802 | 19.96 | 22.903 | 27.21 |
| 184 | 14.848 | 16.182 | 17.853 | 20.022 | 22.975 | 27.288 |
| 185 | 14.882 | 16.224 | 17.904 | 20.082 | 23.046 | 27.365 |
| 186 | 14.916 | 16.265 | 17.954 | 20.143 | 23.116 | 27.441 |
| 187 | 14.95 | 16.306 | 18.004 | 20.203 | 23.186 | 27.515 |
| 188 | 14.982 | 16.347 | 18.053 | 20.262 | 23.255 | 27.59 |
| 189 | 15.015 | 16.387 | 18.103 | 20.321 | 23.324 | 27.662 |
| 190 | 15.047 | 16.427 | 18.151 | 20.38 | 23.391 | 27.734 |
| 191 | 15.078 | 16.466 | 18.199 | 20.438 | 23.459 | 27.805 |
| 192 | 15.109 | 16.505 | 18.247 | 20.495 | 23.525 | 27.875 |
| 193 | 15.14 | 16.543 | 18.295 | 20.552 | 23.591 | 27.943 |
| 194 | 15.17 | 16.581 | 18.342 | 20.608 | 23.656 | 28.011 |
| 195 | 15.199 | 16.619 | 18.388 | 20.664 | 23.721 | 28.078 |
| 196 | 15.228 | 16.656 | 18.434 | 20.72 | 23.785 | 28.143 |
| 197 | 15.257 | 16.692 | 18.479 | 20.774 | 23.847 | 28.207 |
| 198 | 15.285 | 16.728 | 18.524 | 20.829 | 23.91 | 28.271 |
| 199 | 15.312 | 16.763 | 18.568 | 20.882 | 23.972 | 28.334 |
| 200 | 15.339 | 16.798 | 18.612 | 20.936 | 24.032 | 28.395 |
| 201 | 15.365 | 16.833 | 18.655 | 20.988 | 24.093 | 28.456 |
| 202 | 15.391 | 16.867 | 18.698 | 21.04 | 24.152 | 28.515 |
| 203 | 15.417 | 16.9 | 18.741 | 21.091 | 24.211 | 28.573 |
| 204 | 15.441 | 16.933 | 18.782 | 21.142 | 24.269 | 28.63 |
| 205 | 15.465 | 16.965 | 18.823 | 21.192 | 24.327 | 28.687 |
| 206 | 15.489 | 16.997 | 18.864 | 21.242 | 24.383 | 28.742 |
| 207 | 15.512 | 17.028 | 18.904 | 21.291 | 24.439 | 28.797 |
| 208 | 15.534 | 17.059 | 18.944 | 21.34 | 24.494 | 28.85 |
| 209 | 15.556 | 17.089 | 18.983 | 21.388 | 24.549 | 28.903 |
| 210 | 15.577 | 17.118 | 19.022 | 21.435 | 24.603 | 28.954 |
| 211 | 15.598 | 17.147 | 19.06 | 21.482 | 24.656 | 29.005 |
| 212 | 15.618 | 17.176 | 19.097 | 21.528 | 24.708 | 29.054 |
| 213 | 15.637 | 17.204 | 19.134 | 21.574 | 24.76 | 29.103 |
| 214 | 15.656 | 17.231 | 19.171 | 21.619 | 24.811 | 29.15 |

| Month | SD3neg | SD2neg | SD1neg | SD0 | SD1 | SD2 |
|-------|--------|--------|--------|--------|--------|--------|
| 215 | 15.674 | 17.258 | 19.207 | 21.664 | 24.861 | 29.197 |
| 216 | 15.692 | 17.284 | 19.242 | 21.708 | 24.911 | 29.243 |
| 217 | 15.709 | 17.31 | 19.277 | 21.751 | 24.959 | 29.287 |
| 218 | 15.725 | 17.335 | 19.311 | 21.794 | 25.008 | 29.331 |
| 219 | 15.741 | 17.36 | 19.344 | 21.836 | 25.055 | 29.373 |
| 220 | 15.756 | 17.383 | 19.377 | 21.877 | 25.102 | 29.415 |
| 221 | 15.771 | 17.407 | 19.41 | 21.918 | 25.147 | 29.455 |
| 222 | 15.784 | 17.429 | 19.442 | 21.958 | 25.193 | 29.496 |
| 223 | 15.798 | 17.452 | 19.473 | 21.998 | 25.237 | 29.534 |
| 224 | 15.811 | 17.473 | 19.504 | 22.037 | 25.281 | 29.572 |
| 225 | 15.823 | 17.495 | 19.535 | 22.076 | 25.324 | 29.609 |
| 226 | 15.834 | 17.515 | 19.564 | 22.114 | 25.366 | 29.646 |
| 227 | 15.845 | 17.535 | 19.594 | 22.151 | 25.408 | 29.681 |
| 228 | 15.855 | 17.554 | 19.622 | 22.188 | 25.449 | 29.716 |

For non-commercial use only

Table 6-1-4 BMI Classification Criteria for 5-19 Years Old (Female)

| Month | SD3neg | SD2neg | SD1neg | SD0 | SD1 | SD2 |
|-------|--------|---------------|--------|--------|--------|--------|
| 61 | 11.77 | 12.748 | 13.891 | 15.244 | 16.87 | 18.858 |
| 62 | 11.763 | 12.741 | 13.885 | 15.243 | 16.879 | 18.886 |
| 63 | 11.757 | 12.734 | 13.881 | 15.243 | 16.889 | 18.915 |
| 64 | 11.752 | 12.728 | 13.876 | 15.244 | 16.9 | 18.946 |
| 65 | 11.746 | 12.723 | 13.872 | 15.245 | 16.911 | 18.977 |
| 66 | 11.742 | 12.718 | 13.869 | 15.246 | 16.923 | 19.009 |
| 67 | 11.737 | 12.714 | 13.866 | 15.249 | 16.936 | 19.042 |
| 68 | 11.733 | 12.71 | 13.864 | 15.252 | 16.95 | 19.077 |
| 69 | 11.73 | 12.706 | 13.863 | 15.255 | 16.964 | 19.112 |
| 70 | 11.727 | 12.703 | 13.862 | 15.259 | 16.979 | 19.148 |
| 71 | 11.725 | 12.701 | 13.862 | 15.264 | 16.995 | 19.185 |
| 72 | 11.723 | 12.7 | 13.862 | 15.27 | 17.011 | 19.224 |
| 73 | 11.722 | 12.699 | 13.863 | 15.276 | 17.029 | 19.264 |
| 74 | 11.721 | 12.698 | 13.865 | 15.283 | 17.047 | 19.305 |
| 75 | 11.721 | 12.699 | 13.867 | 15.291 | 17.067 | 19.347 |
| 76 | 11.722 | 12.7 | 13.87 | 15.3 | 17.087 | 19.391 |
| 77 | 11.723 | 12.701 | 13.874 | 15.31 | 17.108 | 19.436 |
| 78 | 11.725 | 12.704 | 13.879 | 15.32 | 17.131 | 19.482 |
| 79 | 11.727 | 12.707 | 13.885 | 15.331 | 17.154 | 19.529 |
| 80 | 11.731 | 12.711 | 13.892 | 15.344 | 17.179 | 19.578 |
| 81 | 11.735 | 12.716 | 13.899 | 15.357 | 17.204 | 19.628 |
| 82 | 11.74 | 12.721 | 13.907 | 15.372 | 17.231 | 19.68 |
| 83 | 11.745 | 12.728 | 13.916 | 15.387 | 17.259 | 19.734 |
| 84 | 11.751 | 12.735 | 13.927 | 15.404 | 17.289 | 19.789 |
| 85 | 11.758 | 12.743 | 13.938 | 15.421 | 17.319 | 19.845 |
| 86 | 11.766 | 12.752 | 13.95 | 15.44 | 17.35 | 19.903 |
| 87 | 11.774 | 12.762 | 13.963 | 15.459 | 17.383 | 19.963 |
| 88 | 11.783 | <b>12.772</b> | 13.976 | 15.48 | 17.417 | 20.023 |
| 89 | 11.793 | 12.783 | 13.991 | 15.501 | 17.452 | 20.085 |
| 90 | 11.803 | 12.795 | 14.007 | 15.524 | 17.488 | 20.149 |
| 91 | 11.814 | 12.808 | 14.023 | 15.548 | 17.526 | 20.214 |
| 92 | 11.826 | 12.822 | 14.041 | 15.572 | 17.564 | 20.281 |
| 93 | 11.838 | 12.836 | 14.059 | 15.598 | 17.604 | 20.349 |
| 94 | 11.851 | 12.852 | 14.078 | 15.625 | 17.645 | 20.418 |
| 95 | 11.865 | 12.868 | 14.099 | 15.652 | 17.687 | 20.489 |
| 96 | 11.879 | 12.884 | 14.12 | 15.681 | 17.73 | 20.561 |
| 97 | 11.895 | 12.902 | 14.142 | 15.711 | 17.774 | 20.634 |
| 98 | 11.91 | 12.92 | 14.164 | 15.742 | 17.82 | 20.709 |
| 99 | 11.927 | 12.94 | 14.188 | 15.773 | 17.866 | 20.784 |

| Month | SD3neg | SD2neg | SD1neg | SD0 | SD1 | SD2 |
|-------|--------|--------|--------|--------|--------|--------|
| 100 | 11.944 | 12.959 | 14.212 | 15.806 | 17.914 | 20.862 |
| 101 | 11.962 | 12.98 | 14.238 | 15.839 | 17.962 | 20.94 |
| 102 | 11.98 | 13.001 | 14.264 | 15.874 | 18.012 | 21.019 |
| 103 | 11.998 | 13.023 | 14.291 | 15.909 | 18.062 | 21.1 |
| 104 | 12.018 | 13.045 | 14.318 | 15.945 | 18.113 | 21.181 |
| 105 | 12.037 | 13.068 | 14.346 | 15.982 | 18.166 | 21.263 |
| 106 | 12.057 | 13.092 | 14.375 | 16.019 | 18.219 | 21.346 |
| 107 | 12.078 | 13.115 | 14.404 | 16.058 | 18.272 | 21.429 |
| 108 | 12.099 | 13.14 | 14.434 | 16.096 | 18.326 | 21.513 |
| 109 | 12.12 | 13.165 | 14.465 | 16.136 | 18.381 | 21.599 |
| 110 | 12.141 | 13.19 | 14.496 | 16.176 | 18.437 | 21.684 |
| 111 | 12.163 | 13.216 | 14.527 | 16.217 | 18.493 | 21.77 |
| 112 | 12.185 | 13.242 | 14.559 | 16.258 | 18.551 | 21.857 |
| 113 | 12.208 | 13.269 | 14.592 | 16.3 | 18.608 | 21.944 |
| 114 | 12.231 | 13.296 | 14.625 | 16.343 | 18.666 | 22.031 |
| 115 | 12.254 | 13.323 | 14.659 | 16.386 | 18.725 | 22.12 |
| 116 | 12.278 | 13.352 | 14.694 | 16.43 | 18.785 | 22.208 |
| 117 | 12.302 | 13.38 | 14.729 | 16.475 | 18.846 | 22.298 |
| 118 | 12.327 | 13.41 | 14.764 | 16.52 | 18.907 | 22.388 |
| 119 | 12.352 | 13.439 | 14.801 | 16.566 | 18.969 | 22.479 |
| 120 | 12.378 | 13.47 | 14.838 | 16.613 | 19.032 | 22.57 |
| 121 | 12.404 | 13.501 | 14.876 | 16.661 | 19.096 | 22.663 |
| 122 | 12.43 | 13.533 | 14.914 | 16.71 | 19.161 | 22.755 |
| 123 | 12.458 | 13.565 | 14.954 | 16.76 | 19.226 | 22.849 |
| 124 | 12.485 | 13.598 | 14.994 | 16.81 | 19.293 | 22.943 |
| 125 | 12.514 | 13.631 | 15.035 | 16.861 | 19.36 | 23.038 |
| 126 | 12.542 | 13.666 | 15.076 | 16.914 | 19.429 | 23.134 |
| 127 | 12.572 | 13.7 | 15.119 | 16.967 | 19.498 | 23.231 |
| 128 | 12.602 | 13.736 | 15.162 | 17.021 | 19.568 | 23.328 |
| 129 | 12.632 | 13.772 | 15.206 | 17.076 | 19.639 | 23.426 |
| 130 | 12.663 | 13.81 | 15.251 | 17.132 | 19.712 | 23.525 |
| 131 | 12.695 | 13.847 | 15.297 | 17.188 | 19.785 | 23.624 |
| 132 | 12.727 | 13.885 | 15.343 | 17.246 | 19.859 | 23.725 |
| 133 | 12.76 | 13.925 | 15.39 | 17.304 | 19.933 | 23.825 |
| 134 | 12.793 | 13.964 | 15.438 | 17.364 | 20.009 | 23.927 |
| 135 | 12.827 | 14.004 | 15.487 | 17.424 | 20.086 | 24.029 |
| 136 | 12.861 | 14.045 | 15.536 | 17.485 | 20.163 | 24.131 |
| 137 | 12.896 | 14.087 | 15.586 | 17.546 | 20.241 | 24.234 |
| 138 | 12.931 | 14.129 | 15.637 | 17.609 | 20.32 | 24.338 |
| 139 | 12.967 | 14.171 | 15.688 | 17.672 | 20.4 | 24.442 |

| Month | SD3neg | SD2neg | SD1neg | SD0 | SD1 | SD2 |
|-------|--------|--------|--------|--------|--------|--------|
| 140 | 13.003 | 14.214 | 15.74 | 17.736 | 20.48 | 24.546 |
| 141 | 13.04 | 14.258 | 15.793 | 17.8 | 20.561 | 24.651 |
| 142 | 13.077 | 14.302 | 15.846 | 17.865 | 20.642 | 24.756 |
| 143 | 13.114 | 14.346 | 15.899 | 17.931 | 20.724 | 24.861 |
| 144 | 13.151 | 14.391 | 15.953 | 17.997 | 20.806 | 24.967 |
| 145 | 13.189 | 14.436 | 16.008 | 18.063 | 20.889 | 25.072 |
| 146 | 13.227 | 14.481 | 16.062 | 18.13 | 20.972 | 25.177 |
| 147 | 13.265 | 14.526 | 16.117 | 18.197 | 21.055 | 25.282 |
| 148 | 13.303 | 14.572 | 16.172 | 18.264 | 21.138 | 25.387 |
| 149 | 13.341 | 14.618 | 16.227 | 18.331 | 21.222 | 25.491 |
| 150 | 13.379 | 14.663 | 16.282 | 18.399 | 21.305 | 25.596 |
| 151 | 13.418 | 14.709 | 16.338 | 18.466 | 21.388 | 25.699 |
| 152 | 13.456 | 14.755 | 16.393 | 18.533 | 21.471 | 25.802 |
| 153 | 13.494 | 14.8 | 16.448 | 18.601 | 21.554 | 25.905 |
| 154 | 13.531 | 14.846 | 16.503 | 18.668 | 21.637 | 26.007 |
| 155 | 13.569 | 14.891 | 16.558 | 18.735 | 21.719 | 26.107 |
| 156 | 13.606 | 14.936 | 16.612 | 18.801 | 21.8 | 26.207 |
| 157 | 13.643 | 14.981 | 16.667 | 18.868 | 21.882 | 26.307 |
| 158 | 13.68 | 15.025 | 16.721 | 18.934 | 21.962 | 26.405 |
| 159 | 13.717 | 15.07 | 16.775 | 18.999 | 22.042 | 26.501 |
| 160 | 13.753 | 15.113 | 16.828 | 19.064 | 22.122 | 26.598 |
| 161 | 13.788 | 15.157 | 16.881 | 19.129 | 22.201 | 26.693 |
| 162 | 13.824 | 15.2 | 16.934 | 19.193 | 22.279 | 26.786 |
| 163 | 13.859 | 15.243 | 16.986 | 19.257 | 22.357 | 26.879 |
| 164 | 13.893 | 15.285 | 17.037 | 19.32 | 22.433 | 26.97 |
| 165 | 13.927 | 15.327 | 17.088 | 19.382 | 22.509 | 27.06 |
| 166 | 13.961 | 15.368 | 17.139 | 19.444 | 22.584 | 27.149 |
| 167 | 13.994 | 15.408 | 17.188 | 19.504 | 22.658 | 27.235 |
| 168 | 14.026 | 15.448 | 17.238 | 19.565 | 22.731 | 27.321 |
| 169 | 14.058 | 15.488 | 17.286 | 19.624 | 22.803 | 27.406 |
| 170 | 14.089 | 15.526 | 17.334 | 19.682 | 22.874 | 27.489 |
| 171 | 14.119 | 15.564 | 17.38 | 19.74 | 22.943 | 27.57 |
| 172 | 14.149 | 15.601 | 17.427 | 19.797 | 23.012 | 27.65 |
| 173 | 14.179 | 15.638 | 17.472 | 19.852 | 23.079 | 27.727 |
| 174 | 14.207 | 15.674 | 17.516 | 19.907 | 23.145 | 27.804 |
| 175 | 14.235 | 15.709 | 17.56 | 19.961 | 23.21 | 27.879 |
| 176 | 14.262 | 15.743 | 17.603 | 20.013 | 23.273 | 27.951 |
| 177 | 14.288 | 15.776 | 17.644 | 20.065 | 23.336 | 28.023 |
| 178 | 14.314 | 15.809 | 17.685 | 20.115 | 23.396 | 28.091 |
| 179 | 14.338 | 15.841 | 17.725 | 20.164 | 23.456 | 28.159 |

| Month | SD3neg | SD2neg | SD1neg | SD0 | SD1 | SD2 |
|-------|--------|--------|--------|--------|--------|--------|
| 180 | 14.362 | 15.871 | 17.764 | 20.212 | 23.514 | 28.224 |
| 181 | 14.385 | 15.901 | 17.802 | 20.26 | 23.57 | 28.289 |
| 182 | 14.408 | 15.93 | 17.839 | 20.305 | 23.625 | 28.35 |
| 183 | 14.429 | 15.958 | 17.874 | 20.35 | 23.679 | 28.411 |
| 184 | 14.45 | 15.985 | 17.909 | 20.393 | 23.731 | 28.469 |
| 185 | 14.469 | 16.012 | 17.943 | 20.436 | 23.782 | 28.525 |
| 186 | 14.488 | 16.037 | 17.976 | 20.477 | 23.832 | 28.58 |
| 187 | 14.507 | 16.062 | 18.008 | 20.517 | 23.88 | 28.634 |
| 188 | 14.524 | 16.085 | 18.039 | 20.556 | 23.927 | 28.684 |
| 189 | 14.541 | 16.108 | 18.069 | 20.594 | 23.972 | 28.734 |
| 190 | 14.557 | 16.13 | 18.098 | 20.631 | 24.017 | 28.782 |
| 191 | 14.572 | 16.151 | 18.126 | 20.666 | 24.06 | 28.828 |
| 192 | 14.586 | 16.172 | 18.153 | 20.701 | 24.101 | 28.873 |
| 193 | 14.6 | 16.191 | 18.179 | 20.734 | 24.141 | 28.915 |
| 194 | 14.613 | 16.21 | 18.205 | 20.767 | 24.18 | 28.956 |
| 195 | 14.625 | 16.228 | 18.229 | 20.798 | 24.218 | 28.996 |
| 196 | 14.636 | 16.245 | 18.253 | 20.829 | 24.254 | 29.034 |
| 197 | 14.647 | 16.261 | 18.275 | 20.858 | 24.29 | 29.07 |
| 198 | 14.656 | 16.277 | 18.297 | 20.886 | 24.324 | 29.105 |
| 199 | 14.666 | 16.291 | 18.318 | 20.914 | 24.356 | 29.138 |
| 200 | 14.674 | 16.305 | 18.338 | 20.94 | 24.388 | 29.17 |
| 201 | 14.682 | 16.318 | 18.357 | 20.966 | 24.418 | 29.201 |
| 202 | 14.689 | 16.331 | 18.376 | 20.99 | 24.448 | 29.23 |
| 203 | 14.695 | 16.343 | 18.393 | 21.014 | 24.476 | 29.257 |
| 204 | 14.701 | 16.354 | 18.411 | 21.037 | 24.503 | 29.283 |
| 205 | 14.707 | 16.365 | 18.427 | 21.059 | 24.53 | 29.308 |
| 206 | 14.711 | 16.375 | 18.443 | 21.08 | 24.555 | 29.333 |
| 207 | 14.716 | 16.384 | 18.458 | 21.101 | 24.58 | 29.355 |
| 208 | 14.719 | 16.393 | 18.472 | 21.121 | 24.603 | 29.376 |
| 209 | 14.722 | 16.401 | 18.486 | 21.14 | 24.626 | 29.398 |
| 210 | 14.725 | 16.409 | 18.499 | 21.159 | 24.649 | 29.418 |
| 211 | 14.728 | 16.417 | 18.512 | 21.177 | 24.67 | 29.436 |
| 212 | 14.73 | 16.424 | 18.525 | 21.194 | 24.691 | 29.455 |
| 213 | 14.731 | 16.431 | 18.537 | 21.212 | 24.712 | 29.472 |
| 214 | 14.733 | 16.437 | 18.548 | 21.228 | 24.731 | 29.489 |
| 215 | 14.734 | 16.443 | 18.56 | 21.244 | 24.75 | 29.505 |
| 216 | 14.734 | 16.448 | 18.571 | 21.26 | 24.769 | 29.52 |
| 217 | 14.735 | 16.454 | 18.581 | 21.276 | 24.788 | 29.536 |
| 218 | 14.735 | 16.459 | 18.592 | 21.291 | 24.805 | 29.55 |
| 219 | 14.735 | 16.463 | 18.601 | 21.306 | 24.823 | 29.564 |

| Month | SD3neg | SD2neg | SD1neg | SD0 | SD1 | SD2 |
|-------|--------|--------|--------|--------|--------|--------|
| 220 | 14.734 | 16.468 | 18.611 | 21.32 | 24.84 | 29.577 |
| 221 | 14.734 | 16.473 | 18.621 | 21.334 | 24.856 | 29.589 |
| 222 | 14.733 | 16.477 | 18.63 | 21.348 | 24.873 | 29.602 |
| 223 | 14.732 | 16.48 | 18.639 | 21.362 | 24.889 | 29.614 |
| 224 | 14.731 | 16.484 | 18.648 | 21.375 | 24.905 | 29.626 |
| 225 | 14.729 | 16.488 | 18.657 | 21.388 | 24.92 | 29.637 |
| 226 | 14.728 | 16.491 | 18.665 | 21.401 | 24.935 | 29.649 |
| 227 | 14.726 | 16.494 | 18.673 | 21.414 | 24.951 | 29.659 |
| 228 | 14.724 | 16.497 | 18.681 | 21.427 | 24.965 | 29.67 |

For non-commercial use only

[Leuprorelin-4002] [V3.0] [LK-2021-368] [20250528]

# Appendix B Description of LH and FSH Test Results for Urinary Gn of the First morning void (FMV)

# **Description of Test Results**

Study title: lticenter, Single-arm and Prospective Study to Assess the Efficacy and

Safety of e Treatment of CPP

Client: Lin Beijing) Co., Ltd.

Partner: Ji -Test Med-Tech Co., Ltd.

According of both parties, Jiangsu Macro&Micro-Test Med-Tech Co., Ltd., entrusted by LinkDoc Technology (Beijing) Co., Ltd., conduct tests on luteinizing hormone (LH) and follicle stimulating hormone (FSH) in urine samples in accordance with the criteria of *Collection and Processing of Human Urine Samples* (GB/T38735-2020) in the above study of leuprolide acetate, and issue test reports accordingly. The names of the corresponding detection kits are: Detection Kit for Luteinizing Hormone (LH) (Fluorescent Immunochromatographic Assay), Detection Kit for Follicle Stimulating Hormone (FSH) (Fluorescent Immunochromatographic Assay). See Table 1 for the limit of detection, linear interval and limit of blank range of the kits.

Table 1. Limit of Detection, Linear Interval and Limit of Blank Range of the Lits

| Product name | Limit of detection | Linear interval | Limit of<br>blank | Urine |
|---|---|---|---|---|
| Detection Kit for Luteinizing Hormone (LH)<br>(Fluorescent Immunochromatographic Assay) | 0.05mIU/mL | 0.05-100mIU/mL | 0.02mIU/mL | Urine |
| Detection Kit for Follicle Stimulating Hormone (FSH) (Fluorescent Immunochromatographic Assay) | 0.05mHJ/mL | 0.05~100mIU/mL | 0.02mIU/mL | Urine |
| Detection Kit for Luteinizing Hormone (LH) (Fluorescent Immunochromatographic Assay) | 0.5mIU/mL | 1~100mIU/mL | 1mIU/mL | Blood |
| Detection Kit for Follicle Stimulating Hormone<br>(FSH) (Fluorescent Immunochromatographic<br>Assay) | 0.2mIU/mL | 1-100mIU/mL | 1mIU/mL | Blood |

We recently received feedback from client that the range values of "FSH < 0.2 mIU/mL" and "LH < 0.5 mIU/mL" appeared in the two test reports of 2025.03.10 and 2025.03.14 tests (see Annex 1 Original Report), which are inconsistent with the previous fixed-value test results. For this reason, we have made the following explanations after conducting an internal investigation.

#### 1. Reasons for the range value in the test results.

Our Detection Kit for Luteinizing Hormone (LH) and Follicle Stimulating Hormone (FSH) are used to detect LH and FSH in blood and urine. In previous collaborations with other clients, for test results of blood sample, range values are reported for those below the limit of blank, while fixed values are reported for test results of urine sample.

When we provided the urine sample test for LinkDoc Technology (Beijing) Co., Ltd., the Company also reported fixed values for test results of urine sample in accordance with relevant regulations. However, range results such as <0.2 mIU/mL or <0.5 mIU/mL appeared in the test reports dated March 10, 2025, and March 14, 2025, which was inconsistent with the lowest detection limit of 0.05 mIU/mL shown in the technical document. Because the operator judged the reported result as set as the lower limit of quantification of the test for the blood, the result was reported as the range value. (See Table 2)



| Incorre | ct settings | | Correct settings | | |
|---|---|---|---|---|---|
| Modified conclusion in | n concentration | × | Modified conclusion in reference range | concentration | × |
| | reference range | | | | |
| Name of result | | | Name of result | | |
| determination interval | <0.5mIU/mL | | determination interval | | |
| 1 | | | 1 | | |
| Modified conclusion in | n concentration | × | | | |
| reference range | | ^ | | | |
| Name of result | | | | | |
| determination interval | <0.2mIU/mL | | | | |
| 1 | | | | | |

2. Explanation of the effect of incorrect settings of the judgment interval for the test results reported by the instrument on the test results

The reporting format is realized through the setting of the result judgment interval of the instrument, which will not affect the sample testing process, calculation results, nor the authenticity of the data. As shown in Figure 1 below, the same sample is tested by two report forms and the report is output. If the result judgment interval is set, the range value will be output. If the range interval is not set, the fixed value will be reported.

However, the data issued by our company for 0.05 mIU/mL below the limit of detection are based on the data obtained by reporting the fixed value of urine sample. Although there are specific values for the data, the total error of quantitative detection is greater than 30%, which is of low quantitative significance.

Figure 1 Report Results of the Same Sample by Two Reporting Forms



3. Explanation of Handling for Reports with Range Values.

Based on the explanations in points 1 and 2, for the samples tested on March 10, 2025, and March 14, 2025, we re-output the original results in accordance with the reporting format for urine samples to obtain new result reports (see Appendix 2: Revised Reports). A comparison of the results involving range values in the two reports is shown in Table 3. Both the reports before and after revision, together with this explanation, will be archived in accordance with relevant requirements and delivered to the client for archiving.

Table 3. Original Test Results and Corrected Results of Samples

| Sample | | | | | | | Test Results | | |
|---|---|---|---|---|---|---|---|---|---|
| receivin<br>g<br>hospital | The First Affiliated Hospital, Sun Yat-sen University | | | | | Incorrectly reported results | | Corrected results | |
| Patient No. | Visit<br>numb<br>er | Gender | Abbreviati<br>ons of<br>Pinyin | Lot No. of<br>Reagent | Test<br>date | FSH | LH | FSH | LH |
| | V4 | Female | YWHA | LH | | <0.2mIU<br>/mL | <0.5mIU/<br>mL | 0.07mIU/<br>mL | 0.05mIU/<br>mL |
| | V4 | Female | HURU | FSH | 2025 | 0.95mIU/<br>mL | <0.5mIU/<br>mL | 0.95mIU/<br>mL | 0.04mIU/<br>mL |
| | V3 | Female | PYJL | LH | | <0.2mIU<br>/mL | <0.5mIU/<br>mL | 0.02mIU/<br>mL | 0.03mIU/<br>mL |
| | V3 | Female | WCXI | FSH: | 2025 | <0.2mIU<br>/mL | 4.93mIU/<br>mL | 0.03mIU/<br>mL | 4.93mIU/<br>mL |

Describe herein.

Jiangsu Macro&Micro-Test M

Jiangsu Macro&Micro-Test Med-Tech Co., Ltd.

# **Document History**

| Version<br>No. | Version Date | Author | Major Modifications/Comments |
|---|---|---|---|
| V1.0 | September 21, 2023 | | First version, finalized based on Protocol V3.0. |
| V2.0 | December 6, 2023 | or non-cor | 1.Considering the exposure cycle, an analysis of drug exposure duration is added to the drug exposure status in Section 5.4, with the supplementary calculation formula 2): "Duration of drug exposure (days) = date of last injection of leuprolide for the subject - date of first injection of leuprolide for the subject - date of first injection of leuprolide for the subject + 84". The original serial numbers 2) to 10) of the subsequent calculation formulas are postponed to 3) to 11); the section of drug exposure duration in "Table 6.4.1 Description of Leuprolide Use by Subjects – Enrolled Population" of the corresponding statistical analysis table template is added. 2. Due to the mismatch between the calculation formula and the unit, the original formula 8) in the drug exposure of Section 5.4 is revised as follows: Actual dose used (ug/kg/4w) = Actual dose used (ug/kg)/actual time interval (Month) from current injection to the next injection of leuprolide (Month) = [actual dose used (mg)*1000/body weight (kg)]/[(date of next injection - date of current injection)/30.4375. If there is no next injection, fill in the actual time interval with three months; Revised to: 9) Actual dose used (ug/kg/4w) = Actual dose used (ug/kg)/actual time interval (4w) from current injection to the next injection of leuprolide (4w) = [actual dose used (mg)*1000/body weight (kg)]/[(date of next injection - date of current injection)/28. If there is no next injection - date of current injection)/28. If there is no next injection, fill in the actual time interval with three 4Ws; 3. Add a new Section 5.8 for Analysis of Other Indicators to describe the test results of estradiol/testosterone at each visit and the changes before and after the treatment. Add Section 6.8 of the template of corresponding statistical analysis table, and the numbers of the subsequent sections should be postponed to 6.9, 6.10, and 6.11. |

| Version<br>No. | Version Date | Author | Major Modifications/Comments |
|---|---|---|---|
| V3.0 | May 28, 2025 | of hon-core | 1. Considering the effect of major protocol deviations on data, add handling measures for data affected by major protocol deviations in Section 4 Enrolled Population. Remove "Drug Exposure" from the analysis of the enrolled population and add it to the analysis based on the safety population. 2. Add the drug exposure duration in "Table 6.4.1 Description of Leuprolide Use by Subjects – Enrolled Population" of the statistical analysis table template corresponding to Section 5.4 Drug Exposure. 3. Revise Section 4) of 5.7: LH and FSH results of urinary Gn of in the first morning void (FMV) require programmatic processing before analysis. Additionally, conduct a sensitivity analysis on data directly collected by EDC system, and modify/add corresponding statistical charts accordingly. 4. Add Section 6.8 of the template of statistical analysis table corresponding to Section 5.8 Analysis of Other Indicators. Subsequent section numbers should be adjusted to 6.9, 6.10, and 6.11. 5. Given the refinement of the enrolled population definition and the imputation of missing values for some time variables in this SAP, add Section 5.13 to explain inconsistencies between the SAP and the Study Protocol. 6. Revise the BMI grading criteria in Section 5.3 and update the information in Appendix B. 7. According to the Protocol, the primary endpoint should display trend changes by visits and genders. Therefore, in sections related to LH suppression in the GnRH stimulation test (e.g., Sections 5.6 and 5.10), add an analysis of LH suppression achieved at Week 12 of the visit in the GnRH stimulation test. 8. Add the list of results corresponding to Sections 5.6, 5.7 and 5.8. 9. Delete original Appendix A, and calculate the predicted adult height using the BP method. After evaluation by the project team and Investigators, this method is found to overestimate adult height and is deemed unsuitable for this study. The project team recommend using the formula developed "based on BP method principles combined with the survey data of nin |

Note: Compared with the Chinese version, the dictionary version in the English SAP has been updated according to the latest actual situation.

#### References

- [1] WHO. Growth reference data for 5-19 years. <a href="https://www.who.int/tools/growth-reference-data-for-5to19-years/indicators/bmi-for-age">https://www.who.int/tools/growth-reference-data-for-5to19-years/indicators/bmi-for-age</a>.
- [2] Liang Yan, Wei Hong, Yu Xiao, Song Ningyi, Luo Xiaoping. Application of a New Height Prediction Method in the Treatment of Girls with Idiopathic Central Precocious Puberty with Gonadotropin-releasing hormone analogs [J]. Chinese Journal of Pediatrics, 2015,53(11):840-844.
- [3] Li Hui, Ji Chengye, Zong Xinnan, Zhang Yaqin. Standardized Growth Curve of Height and Weight of Children and Adolescents Aged 0-18 Years in China [J]. Chinese Journal of Pediatrics, 2009, 47(7):487-492.

For non-commercial use only